CLINICAL TRIAL: NCT07348900
Title: The Effect of Recreational Play Activities on Anxiety Levels of Children Undergoing Chemotherapy and Their Parents: A Quasi-Experimental Study
Brief Title: Effect of Recreational Play Activities on Anxiety in Children Receiving Chemotherapy and Their Parents
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sule ŞENOL, PhD, Akdeniz University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 241; 241 (Registry Identifier: University Clinical Research Ethics Committee (Turkey))
Record Dates: First submitted 2026-01-09; First posted 2026-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Anxiety; Pain
Keywords: Pediatric Oncology; Chemotherapy; Play-based Intervention; Parents; Anxiety
MeSH Terms: conditions — Anxiety Disorders; Pain

STUDY DESIGN:
Intervention Model Description: This quasi-experimental study used a single-group pretest-posttest design. Participants received structured play-based supportive care activities in addition to routine care, and outcomes were assessed before and after the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Play-Based Intervention Group (Experimental): Children and their parents received structured play-based supportive care activities in addition to routine chemotherapy care.
  Interventions: Behavioral: Play-Based Supportive Care Activities

INTERVENTIONS:
Behavioral: Play-Based Supportive Care Activities — Structured play-based supportive care activities were provided to children during chemotherapy sessions to reduce anxiety and pain and to support emotional coping. Parents accompanied the children during the activities.

SUMMARY:
Children receiving chemotherapy often experience high levels of anxiety, which may also affect their parents. Anxiety during treatment can negatively influence emotional well-being, treatment adherence, and overall quality of life. Non-pharmacological and supportive interventions, such as recreational play activities, may help reduce anxiety in pediatric patients and their caregivers.

The aim of this study is to evaluate the effect of recreational play activities on anxiety levels of children undergoing chemotherapy and their parents. The study was conducted using a quasi-experimental design in a pediatric oncology setting. Children receiving chemotherapy and their parents participated in structured recreational play activities in addition to routine care. Anxiety levels of both children and parents were assessed before and after the intervention using validated anxiety assessment tools.

The findings of this study are expected to contribute to evidence-based nursing practices by highlighting the potential benefits of recreational play activities as a supportive intervention to reduce anxiety in pediatric oncology patients and their parents.

DETAILED DESCRIPTION:
This study aimed to examine the effect of recreational play activities on anxiety levels of children undergoing chemotherapy and their parents. A quasi-experimental study design was used. The study was conducted in a pediatric oncology unit and included children receiving chemotherapy and their parents who met the inclusion criteria.

Participants were assigned to an intervention group that received structured recreational play activities in addition to routine care. Recreational play activities were planned according to the age and developmental level of the children and were implemented during chemotherapy sessions. The activities included age-appropriate games and play-based interactions designed to promote relaxation, emotional expression, and coping.

Anxiety levels of children and parents were assessed before and after the intervention using validated anxiety measurement scales. Demographic and clinical data were also collected. The primary outcome of the study was the change in anxiety levels of children and parents following participation in recreational play activities.

Ethical approval was obtained from the relevant Clinical Research Ethics Committee prior to the initiation of the study. Written informed consent was obtained from parents, and assent was obtained from children when appropriate. All study procedures were conducted in accordance with ethical principles and institutional guidelines.

The results of this study provide evidence on the effectiveness of recreational play activities as a non-pharmacological nursing intervention to reduce anxiety in pediatric oncology settings and support the integration of play-based approaches into routine clinical care.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 4-10 years receiving inpatient chemotherapy treatment in a pediatric oncology and hematology clinic;
* Children and parents who agreed to participate in the study and provided written informed consent;
* Children able to communicate verbally; parents who are able to read and write in Turkish.

Exclusion Criteria:

* Children who experienced a significant life event unrelated to the disease within the last six months (such as parental divorce, death of a parent, or relocation);
* Children receiving more than one chemotherapy cycle simultaneously;
* Children in the terminal stage of the disease;
* Children or parents who declined participation or withdrew before completion of the study.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 62 (Actual)
Dates: Start 2024-11-15 (Actual); Primary Completion 2025-05-07 (Actual); Study Completion 2025-05-07 (Actual)

PRIMARY OUTCOMES:
Anxiety level of children undergoing chemotherapy | Baseline (before the intervention) and immediately after the intervention during the chemotherapy session
  Children's anxiety was assessed using the Child Anxiety Scale-State (CAS-State), an age-appropriate visual analog scale designed for children aged 4-10 years. The scale ranges from 0 to 10, where higher scores indicate higher levels of state anxiety. Anxiety scores were recorded at baseline (before the play-based recreational activity intervention) and immediately after the intervention during the chemotherapy session.

SECONDARY OUTCOMES:
Parental anxiety level | Baseline (before the intervention) and immediately after the intervention during the chemotherapy session
  Parental anxiety was assessed using the State Anxiety Inventory (STAI-I), a validated self-report questionnaire consisting of 20 items with total scores ranging from 20 to 80, where higher scores indicate higher levels of anxiety.

CONTACTS AND LOCATIONS:
Overall Officials: Şule Şenol, PhD, Principal Investigator — Akdeniz Üniversitesi Hemşirelik Fakültesi
Locations (1):
- Akdeniz University Hospital, Pediatric Oncology and Hematology Clinic, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to the inclusion of pediatric participants and the absence of specific consent for data sharing.